CLINICAL TRIAL: NCT04103112
Title: Compression Hosiery to Avoid Post-Thrombotic Syndrome (CHAPS)
Brief Title: Compression Hosiery to Avoid Post-Thrombotic Syndrome
Acronym: CHAPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the request of the study's funders (NIHR-HTA) the study was terminated early due to poor recruitment in the context of the COVID-19 pandemic and unprecedented pressures faced by the NHS.
Sponsor: Imperial College London (Other)
Collaborators: University of Edinburgh (Other); Universidad de Granada (Other); University College, London (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19CX5434
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-07

CONDITIONS: Deep Vein Thrombosis; Deep Vein Thrombosis Leg; Post Thrombotic Syndrome
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent researcher at each site will perform leg assessments blind to participant allocation. This researcher will not have been involved in recruitment, stocking provision, adherence monitoring or behavioural interventions. Participants will be encouraged to remove their stockings on the day prior to their clinic visit, they will be asked not to discuss the stockings with the independent assessor. Blinding will be assessed by asking the assessors whether the patient attended study visits wearing a stocking, and whether the patient made it known that they had been wearing a stocking or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical care (No Intervention): Standard clinical care (anticoagulation) with no graduated compression stocking
- Graduated compression stocking and standard clinical care (Experimental): A graduated compression stocking and the standard clinical care (anticoagulation)
  Interventions: Device: Graduated compression stocking

INTERVENTIONS:
Device: Graduated compression stocking — Compression stockings have been used safely in the UK for about 50 years. They contain an elastic fibre designed to fit tightly around the legs. These specialist stockings are tighter around the ankle, with the level of compression gradually decreasing up the garment.
  The pressure created by the stockings helps blood flow up the leg, allowing blood to flow freely to the heart and not pool in the leg which can result in pain and swelling.
  Arms: Graduated compression stocking and standard clinical care

SUMMARY:
Patients with a deep vein thrombosis (DVT) may develop long-term symptoms, e.g. lifelong leg pain, skin changes and occasionally ulceration, known as post-thrombotic syndrome (PTS). This affects about half of people with a history of DVT.

This randomised study aims to show whether the regular use of a compression stocking after DVT in the leg, prevents long-term pain, swelling and ulceration. Currently small trials show varied results and a large trial is required to answer the question.

DETAILED DESCRIPTION:
Every year 1 in 1000 persons in the United Kingdom are diagnosed with a blood clot in the leg veins (deep vein thrombosis). In just under half of those with deep vein thrombosis, leg pain, swelling and skin breakdown (ulcers) can occur, a lifelong condition called post-thrombotic syndrome. This impacts upon a person's ability to work, their confidence and independence. In most patients there is no effective treatment and they lose income from unemployment. Ulcers, if they occur, require bandaging that needs to be changed twice weekly.

Treatment guidelines for deep vein thrombosis do not currently include the use of a compression stockings. They can sometimes be difficult to put on for those who cannot bend down, the stockings can slip or roll down, or become uncomfortable in hot weather. Stockings cost the National Health Service (NHS) approximately £50 every 6 months. The evidence for stockings comes from two early trials comparing patients wearing a stocking to those who did not.

There was a large benefit in both these trials for wearing a stocking, with no major side effects. In 2014, a Canadian group published a trial comparing wearing a compression stocking to wearing a non-compressive stocking. The rates of post-thrombotic syndrome were identical. The Canadian trial also suggested that only half of patients actually wear stockings, one reason the trial may have shown no difference. The Canadian trial suggested that stockings did not prevent future thrombosis or help leg pain. Whilst United Kingdom National Institute for Health and Care Excellence (NICE) recommendations are to avoid stockings after deep vein thrombosis, European recommendations are to still wear them. The contradictory results of these three trials have led us to design the CHAPS trial.

The aim of CHAPS is to confirm whether there is a real benefit of wearing stockings in addition to the standard treatment for deep vein thrombosis, which is blood thinning medication.

Adults with a first deep vein thrombosis can join the trial. They will be randomly allocated to receive either blood thinning medication, or blood thinning medication and an additional compression stocking. This is a tight, custom fitted stocking that they will be asked to wear whilst they are awake as much as possible for between 6-30 months. Patients will be aware of which group they are in, but will be asked not to wear the stocking when they come for their assessment. This keeps the researchers impartial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic presentation of first deep vein thrombosis, <2 weeks from diagnosis
* Imaging confirmed, lower limb deep vein thrombosis (popliteal, femoral, iliac or combination)
* Ability to give informed consent
* Age 18 or over

Exclusion Criteria:

* Life expectancy < 2 years
* Contraindication to wearing graduated compression stockings
* Previously intolerant of or already wearing graduated compression stockings for more than 1 month.
* Ankle brachial pressure index (ABPI) <0.8 or pedal pulses absent
* Bilateral deep vein thrombosis
* Previous chronic venous insufficiency (patients with existing chronic skin changes or ulceration, defined as C4,5,6 by Clinical Etiological Anatomical Pathophysiological (CEAP) classification)
* Pre-existing post thrombotic syndrome, significant leg pain (e.g. knee arthritis, spinal claudication) or oedema (e.g. lymphoedema).
* Newly diagnosed cancer, metastatic cancer, or cancer undergoing active treatment or palliation
* Contraindication to anticoagulation
* Known allergy to fabric in compression stockings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Principal Investigator — Imperial College London
Locations (12):
- United Kingdom (12):
  - Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Imperial College Healthcare NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - London North West University Healthcare NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - East Cheshire NHS Trust, Macclesfield
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford
  - Salisbury Hospital NHS Foundation Trust, Salisbury

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Graduated Compression Stocking and Standard Clinical Care: A graduated compression stocking and the standard clinical care (anticoagulation)
  Graduated compression stocking: Compression stockings have been used safely in the UK for about 50 years. They contain an elastic fibre designed to fit tightly around the legs. These specialist stockings are tighter around the ankle, with the level of compression gradually decreasing up the garment.
  The pressure created by the stockings helps blood flow up the leg, allowing blood to flow freely to the heart and not pool in the leg which can result in pain and swelling.
Period: Overall Study
Arm/Group | Standard Clinical Care | Graduated Compression Stocking and Standard Clinical Care
Started | 76 | 76
Completed | 55 | 56
Not Completed | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Clinical Care | Graduated Compression Stocking and Standard Clinical Care | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (14.2) | 56.2 (14.8) | 57.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 29 | 49
  Male | 56 | 47 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 58 | 124
  Mixed Race/Multiple Ethnic Background | 2 | 1 | 3
  Asian or Asian British | 2 | 8 | 10
  Black or Black British | 3 | 6 | 9
  Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post Thrombotic Syndrome (PTS)
Description: Measured using the validated Villalta criteria
Time Frame: 30 months
Measure: Number; unit: Number of PTS events
Arm/Group | Standard Clinical Care | Graduated Compression Stocking and Standard Clinical Care
Number analyzed (Participants) | 55 | 56
Number of PTS events
  Index-Leg | 28 | 17
  Non-Index-Leg | 6 | 9

2. Secondary Outcome: Venous Ulceration Incidence
Description: Measured using the validated Villalta criteria
Time Frame: 30 months
Reporting Status: Not Posted

3. Secondary Outcome: Employment Status
Description: Change in number of days working from baseline
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Clinical Care | Graduated Compression Stocking and Standard Clinical Care
Number analyzed (Participants) | 76 | 76
Participants
  Full time | 34 | 34
  Part time | 8 | 9
  Unemployed | 7 | 5
  Retired | 26 | 27
  Student | 1 | 0
  Missing | 0 | 1

4. Secondary Outcome: Change in Disease-specific and Generic Quality of Life
Description: Measured using VEINES-QoL scale (instrument to measure quality of life in deep venous thrombosis). Two summary scores can be computed. The VEINES-QOL summary score (25 items) provides an estimate of the overall impact of deep venous thrombosis on the patient's quality of life. The VEINES-Sym summary score (10 items) measures symptom severity. Higher scores indicate better outcomes.
Time Frame: 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Disease-specific and Generic Quality of Life
Description: Measured using EuroQoL EQ5D scale (European Quality of Life 5D instrument for measuring generic health status) . A health index on a score of 0 to 1 and the participants' self-rated health on a vertical score of zero to 100. Higher scores indicate better quality of life.
Time Frame: 18 months
Reporting Status: Not Posted

6. Secondary Outcome: The Proportion of Participants Who Are Adherent to Stockings and Anticoagulants
Description: Patient self-report - at six months median follow up, the criteria for continuing CHAPS is equal to or over 70% of participants wearing stockings (monthly self-reported patient adherence questionnaire) for equal to or over 4 days per week in the intervention arm, along with a documented reorder of stockings within the last 6 months.
Time Frame: 30 months
Reporting Status: Not Posted

7. Secondary Outcome: Cost-effectiveness of Stocking Prescription
Description: Incremental cost-effectiveness ratio (ICER) from the EQ-5D questionnaire, with appropriate sensitivity analysis
Time Frame: 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through participant's study completion, 6-30 months (median 18 months)
Arm/Group | Standard Clinical Care | Graduated Compression Stocking and Standard Clinical Care
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 5/76 | 2/76
Other Adverse Events (participants affected / at risk) | 5/76 | 6/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Clinical Care (N=76) | Graduated Compression Stocking and Standard Clinical Care (N=76)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Left posterior Stroke; PE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute MCA infarction (Nervous system disorders) | 1 | 0
Admitted with nose bleed and pr bleed; rectal ca with mets - on palliative chemotherapy (Blood and lymphatic system disorders) | 1 | 0
Pr bleeding, thrombocytopaenia (Blood and lymphatic system disorders) | 1 | 0
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness, collapse, black stools, lack of appetite (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Clinical Care (N=76) | Graduated Compression Stocking and Standard Clinical Care (N=76)
Varicose veins (Vascular disorders) | 1 | 0
Edema (Vascular disorders) | 1 | 0
Gout flare-ups increased in severity since taking warfarin; patient noted an increase in pain (Metabolism and nutrition disorders) | 1 | 0
Leg pain and swelling to left leg. (Vascular disorders) | 1 | 0
Discomfort of fifth toe (Musculoskeletal and connective tissue disorders) | 0 | 1
Indentation from stocking (Musculoskeletal and connective tissue disorders) | 0 | 1
Soreness medial aspect of the shin (Musculoskeletal and connective tissue disorders) | 0 | 1
Pins and needles at the end of first full day of wearing stockings (Nervous system disorders) | 0 | 1
Bruising to leg (Musculoskeletal and connective tissue disorders) | 0 | 1
Patient seen by vascular team and advised to wear class II hoisery (Vascular disorders) | 1 | 0
Acute & chronic DVT of left leg (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT04103112/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT04103112/SAP_001.pdf